CLINICAL TRIAL: NCT06130046
Title: MR-proADM as a Early Biomarker for DGF and AR in Kidney and Liver Transplantation
Acronym: DARE
Status: Recruiting | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Roberta Angelico, Associate Professor, MD, PhD, FEBS, University of Rome Tor Vergata
Other Study IDs: DARE
Record Dates: First submitted 2023-10-12; First posted 2023-11-13 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Kidney Transplant; Complications; Liver Transplant; Complications
Keywords: MR-proADM; Adrenomedullin; Kidney Transplantation; Liver Transplantation; DGF; Acute rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — EDTA Blood Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- OLT: Observation of MR-proADM levels at protocol timepoints to predict main (DGF and AR) and secondary (surgical complications, infections, others) complications after liver transplantation at our Institution.
  Interventions: Biological: MR-proADM dosage
- KT: Observation of MR-proADM levels at protocol timepoints to predict main (DGF and AR) and secondary (surgical complications, urological complications, infections, others) complications after kidney transplantation at our Institution.
  Interventions: Biological: MR-proADM dosage

INTERVENTIONS:
Biological: MR-proADM dosage — Dosage of MR proADM at OLT/KT, 1, 3, 5, 15 POD and 1, 3, 6, 9, 12 months F-U

SUMMARY:
To define the sensibility and the specificity of increased levels of MR-proADM for early, non-invasive, diagnosis of AR and DGF after kidney and liver transplantation creating a predictive model for related complications after kidney and liver transplantation based on the pre-operative and post-operative levels of MR-proADM and by a machine learning process.

DETAILED DESCRIPTION:
Despite long-term outcomes of kidney and liver transplantation significantly improved in the last decades, high morbidity and mortality is still an issue at short term after transplantation. Specifically, occurrence of delayed graft function (DGF) and early acute rejection (AR) may cause multi-organ failure or graft failure, admission to intensive care unit, prolonged hospitalization and high-dosage immunosuppressive therapy which might expose patients to several further complications such as infections, neoplasm, and metabolic disease. Consequently, solid organ transplant recipients represent a very frail population at high risk of complications. Therefore, development of new biomarkers for the prevention and early diagnosis of the major post-transplant complications influencing the morbidity and mortality of solid organ transplant recipients are needed. Adrenomedullin (ADM) is a 52-amino acid peptide with a variety of physiologic functions such as immunemodulating activity, direct bactericidal activity, maintenance of renal homeostasis, and vasodilatory activity. Recent study has shown that midregional proADM (MR-proADM) is co-synthesized with ADM in equimolar amounts and has the advantages of a longer half-life, lack of bioactivity and lack of protein binding. MR-proADM has been recognized as a prognostic marker, stratifying the mortality risk in patients with sepsis in intensive care units. Moreover, recently MD-proADM has been also associated with risk of specific organ failure such as acute kidney injury, acute liver damage, acute respiratory distress syndrome and acute cardiac injury. Literature results suggest that recovery of graft function after KT may lead to decrease in plasma MR-proADM level in patients with ESRD, and that plasma MR-proADM level may could increase in the early phases of DGF and AR after KT and LT as a response damage and to the immune activation. The study will allow to evaluate the utility MR-proADM as an early biomarker of DGF and AR in patients undergoing kidney and liver transplantation at our Institution. Also, the study aims to analyze how the value of this biomarker can change in association with post-transplant complication and to create a predicting model by machine cut-off values of references for MR-proADM.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipient at our Institution
* Liver transplant recipient at our Institution

Exclusion Criteria:

* Re-transplantation
* Dual kidney transplantation
* Combined transplant (kidney-liver, kidney-pancreas)
* Autoimmune disease as indication to transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult kidney or liver transplant recipients who underwent OLT or KT at the University of Rome Tor Vergata with no indication for autoimmune diseases or for combined/dual transplant or re-transplantation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of MR-proADM as biomarker of DGF and AR in OLT/KT | 3 years
  To define the sensibility and the specificity of increased levels of MR-proADM for early, non-invasive, diagnosis of AR and DGF after kidney and liver transplantation.

SECONDARY OUTCOMES:
Accuracy of MR-proAMD for early detection of other complications in OLT/KT | 3 years
  Creating a predictive model of complications after kidney and liver transplantation based on the pre-operative and post-operative levels of MR-proADM by machine learning process.
Algorithm for risk prediction | 3 years
  Development of a software algorithm predicting the risk of post-transplant complications
Digital Pathology Dataset | 3 years
  Development of digital pathology for graft biopsy
MR-proADM Online Dataset | 3 years
  Development of an online platform to collect and correlate data on post-transplant biopsy and MRPro-ADM levels.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Angelico, PhD FEBS, Principal Investigator — University of Rome Tor Vergata
Locations (1):
- University of Rome Tor Vergata, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Legramante JM, Mastropasqua M, Susi B, Porzio O, Mazza M, Miranda Agrippino G, D Agostini C, Brandi A, Giovagnoli G, Di Lecce VN, Bernardini S, Minieri M. Prognostic performance of MR-pro-adrenomedullin in patients with community acquired pneumonia in the Emergency Department compared to clinical severity scores PSI and CURB. PLoS One. 2017 Nov 21;12(11):e0187702. doi: 10.1371/journal.pone.0187702. eCollection 2017. PMID 29161297
- [Background] Minieri M, Di Lecce VN, Lia MS, Maurici M, Bernardini S, Legramante JM. Role of MR-proADM in the risk stratification of COVID-19 patients assessed at the triage of the Emergency Department. Crit Care. 2021 Nov 26;25(1):407. doi: 10.1186/s13054-021-03834-9. No abstract available. PMID 34836547
- [Background] Manzia TM, Lai Q, Hartog H, Aijtink V, Pellicciaro M, Angelico R, Gazia C, Polak WG, Rossi M, Tisone G. Graft weight integration in the early allograft dysfunction formula improves the prediction of early graft loss after liver transplantation. Updates Surg. 2022 Aug;74(4):1307-1316. doi: 10.1007/s13304-022-01270-0. Epub 2022 Mar 19. PMID 35306614
- [Background] Angelico R, Gerlach UA, Gunson BK, Neil D, Mergental H, Isaac J, Muiesan P, Mirza D, Perera MTP. Severe Unresolved Cholestasis Due to Unknown Etiology Leading to Early Allograft Failure Within the First 3 Months of Liver Transplantation. Transplantation. 2018 Aug;102(8):1307-1315. doi: 10.1097/TP.0000000000002139. PMID 29470351
- [Background] Marutsuka K, Nawa Y, Asada Y, Hara S, Kitamura K, Eto T, Sumiyoshi A. Adrenomedullin and proadrenomudullin N-terminal 20 peptide (PAMP) are present in human colonic epithelia and exert an antimicrobial effect. Exp Physiol. 2001 Sep;86(5):543-5. doi: 10.1113/eph8602250. PMID 11571480
- [Background] Minamino N, Kikumoto K, Isumi Y. Regulation of adrenomedullin expression and release. Microsc Res Tech. 2002 Apr 1;57(1):28-39. doi: 10.1002/jemt.10048. PMID 11921354
- [Background] Kita T, Kitamura K. Translational studies of adrenomedullin and related peptides regarding cardiovascular diseases. Hypertens Res. 2022 Mar;45(3):389-400. doi: 10.1038/s41440-021-00806-y. Epub 2022 Jan 6. PMID 34992239
- [Background] Ueda S, Nishio K, Minamino N, Kubo A, Akai Y, Kangawa K, Matsuo H, Fujimura Y, Yoshioka A, Masui K, Doi N, Murao Y, Miyamoto S. Increased plasma levels of adrenomedullin in patients with systemic inflammatory response syndrome. Am J Respir Crit Care Med. 1999 Jul;160(1):132-6. doi: 10.1164/ajrccm.160.1.9810006. PMID 10390390
- [Background] Eto T, Kitamura K. Adrenomedullin and its role in renal diseases. Nephron. 2001 Oct;89(2):121-34. doi: 10.1159/000046059. No abstract available. PMID 11549894
- [Background] Suzuki Y, Itoh H, Katagiri F, Sato F, Kawasaki K, Sato Y, Sato Y, Mimata H, Takeyama M. Relationship between plasma mid-regional pro-adrenomedullin level and resistance to antihypertensive therapy in stable kidney transplant recipients. Peptides. 2013 Oct;48:45-8. doi: 10.1016/j.peptides.2013.08.001. Epub 2013 Aug 13. PMID 23954711
- [Background] Reuken PA, Kiehntopf M, Stallmach A, Bruns T. Mid-regional pro-adrenomedullin (MR-proADM): an even better prognostic biomarker than C-reactive protein to predict short-term survival in patients with decompensated cirrhosis at risk of infection? J Hepatol. 2012 Nov;57(5):1156-8; author reply 1158-9. doi: 10.1016/j.jhep.2012.06.036. Epub 2012 Aug 11. No abstract available. PMID 22892248
- [Background] Valenzuela-Sanchez F, Valenzuela-Mendez B, Rodriguez-Gutierrez JF, Estella-Garcia A, Gonzalez-Garcia MA. New role of biomarkers: mid-regional pro-adrenomedullin, the biomarker of organ failure. Ann Transl Med. 2016 Sep;4(17):329. doi: 10.21037/atm.2016.08.65. PMID 27713887